CLINICAL TRIAL: NCT03478449
Title: A Single Center Randomized Prospective Study on the Criteria for Lymph Node Sorting for Pathological Examination After Curative Surgery for Gastric Cancer
Brief Title: The Criteria for Lymph Node Sorting for Pathological Examination in Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DJY001
Record Dates: First submitted 2018-02-10; First posted 2018-03-27 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Lymph Node Metastases; Gastric Cancer; Exanimation
MeSH Terms: conditions — Lymphatic Metastasis; Stomach Neoplasms; Coma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fine sorting lymph node group (Experimental)
  Interventions: Procedure: lymph node sorting for pathological examination
- Regional sorting lymph node group (No Intervention)

INTERVENTIONS:
Procedure: lymph node sorting for pathological examination — In this study, intervention methods include two kinds of lymph node sorting for pathological examination in gastric cancer samples after curative surgery. One is the fine sorting lymph nodes, representing the lymph nodes should be sorted one by one from the tissues around the stomach, celiac axis, and the main brunches of celiac axis. The other is the group sorting lymph nodes, representing the lymph nodes should be simply sorted in the soft tissues around the stomach, celiac axis, and the main brunches of celiac axis.
  Arms: Fine sorting lymph node group

SUMMARY:
The aim of this study is intending to provide the optimal procedures of lymph node sorting for pathological examination after curative surgery for gastric cancer, which can discriminate the differences of the status of lymph node metastasis, pTNM classification and prognostic outcome of gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Physical conditions compliance with the requirements for curative gastrectomy
* 2) Consent to undergo the D2 lymphadenectomy
* 3) Comply with the protocol during the whole study period
* 4) No neoadjuvant therapy administration
* 5) Sign informed consent and permission of withdraw in the whole study period
* 6) Consent to provide the tissue specimens after surgery for this study
* 7) Pathological examination confirmation the adenocarcinoma of stomach before surgery
* 8) Estimation the overall survival after surgery no less than 6 months
* 9) No anesthesia or operation contraindication disease
* 10) cTanyNanyM0 stage demonstration by CT and endoscopic ultrasonography examinations
* 11) Negative cytological detection in operation
* 12) No seriously concomitance's diseases
* 13) Karnofsky Performance Scores (KPS) more than 60

Exclusion Criteria:

* 1) Women during pregnant stage and breast-feed stage
* 2) Women of childbearing age without any contraceptive measures
* 3) Severe congestive heart failure, frequent arrhythmia, or myocardial infarction within 12 months
* 4) Immunosuppressive therapists for organ transplantation
* 5) Seriously uncontrolled recurrent infection
* 6) other malignant tumors
* 7) No abilities of self-knowledge or mental disorders
* 8) Participating in other clinical trials
* 9) Siewert I and II esophagogastric junction tumors
* 10) Serious internal diseases obstruction surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Migration of pN stage in gastric cancer patients | 60 months
  According to the overall survival of all included patients, we will evaluate the optimal lymph node sorting method to obtain the accurately pathological stage of lymph node metastatic counts (pN stage) for prediction the prognosis of patients after curative surgery for gastric cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03478449/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03478449/SAP_001.pdf
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03478449/ICF_002.pdf